CLINICAL TRIAL: NCT00002631
Title: A PHASE III INTERGROUP RANDOMIZED COMPARISON OF COMBINED MODALITY THERAPY FOR CARCINOMA OF THE ESOPHAGUS: HIGH-DOSE VS CONVENTIONAL-DOSE RADIATION THERAPY
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Cancer of the Esophagus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: RTOG-9405; CDR0000064043; E-R9405; NCCTG-914051; INT-0123
Record Dates: First submitted 1999-11-01; First posted 2004-08-31 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Esophageal Cancer
Keywords: stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Drug Therapy; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: chemotherapy
Drug: cisplatin
Drug: fluorouracil
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not known whether high-dose radiation therapy is more effective than standard dose radiation therapy in treating cancer of the esophagus.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy plus high- or standard-dose radiation therapy in treating patients with cancer of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare, using a prospective controlled randomized study design, the survival and failure patterns associated with conventional-dose radiotherapy and fluorouracil/cisplatin (5-FU/CDDP) vs. high-dose radiotherapy and 5-FU/CDDP in patients with esophageal cancer. II. Compare the tolerance and quality of life of patients receiving these therapies.

OUTLINE: Randomized study. Arm I: Radiotherapy plus 2-Drug Combination Chemotherapy/Radiosensitization. Tumor irradiation using megavoltage photons of at least 6 MV (electrons may be used if required to boost supraclavicular fossa dose); plus Cisplatin, CDDP, NSC-119875; Fluorouracil, 5-FU, NSC-19893. High-dose radiotherapy. Arm II: Radiotherapy plus 2-Drug Combination Chemotherapy/Radiosensitization. Tumor irradiation as in Arm I; plus CDDP/5-FU. Conventional-dose radiotherapy.

PROJECTED ACCRUAL: Up to 298 patients will be entered over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven primary squamous cell or adenocarcinoma of the esophagus Clinical Stage T1-4, Nx, M0 disease required Disease entirely confined to the esophagus and periesophageal soft tissue with no tumor extension within 2 cm proximal to the stomach No biopsy-proven invasion of the tracheal-bronchial tree or tracheal-esophageal (TE) fistula Bronchoscopy of tracheal-bronchial tree required for lesions less than 30 cm from the incisors to exclude TE fistula Negative liver biopsy required if liver CT suggestive of metastatic disease Negative biopsy required for enlarged (1.5 cm or greater) retroperitoneal or celiac nodes seen on CT Negative biopsy of clinically or radiographically positive supraclavicular nodes required with cervical primaries No recurrent disease No multiple carcinomas of the esophagus

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60%-100% Hematopoietic: WBC at least 4,000 Platelets at least 150,000 Hb at least 10 g/dL Hepatic: Not specified Renal: Creatinine normal OR Creatinine clearance at least 65 mL/min Nutrition: Recommended oral intake requirements (by mouth or tube feeding): More than 1.5 x Basal Energy Expenditure (BEE) measured by Harris- Benedict equation OR More than 1,000 calories/sqm of body surface area (BSA) Intravenous hyperalimentation (recommended if inadequate oral intake): 1.75-2.25 x BEE OR 1,200-1,600 calories/sqm BSA Upper limits may be waived for hypermetabolic patients Other: No second malignancy within 5 years except: Curable nonmelanomatous skin cancer Cervical cancer in situ No pregnant or nursing women

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior or concurrent growth factor administration Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior chest irradiation Surgery: No prior resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 1995-06; Primary Completion 1999-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D. Minsky, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Thomas M. Pisansky, MD, Study Chair — Mayo Clinic; James A. Martenson, MD, Study Chair — Mayo Clinic
Locations (18):
- United States (17):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
- Saskatchewan Cancer Agency, Regina, Saskatchewan, Canada

REFERENCES:
- [Background] Thomas CR Jr, Berkey BA, Minsky BD, Gaspar LE, Herskovic A, Rich TA, Gunderson LL. Recursive partitioning analysis of pretreatment variables of 416 patients with locoregional esophageal cancer treated with definitive concomitant chemoradiotherapy on Intergroup and Radiation Therapy Oncology Group trials. Int J Radiat Oncol Biol Phys. 2004 Apr 1;58(5):1405-10. doi: 10.1016/j.ijrobp.2003.09.022. PMID 15050316
- [Background] Smalley SR, Gunderson L, Tepper J, Martenson JA Jr, Minsky B, Willett C, Rich T. Gastric surgical adjuvant radiotherapy consensus report: rationale and treatment implementation. Int J Radiat Oncol Biol Phys. 2002 Feb 1;52(2):283-93. doi: 10.1016/s0360-3016(01)02646-3. PMID 11872272
- [Result] Kachnic LA, Winter K, Wasserman T, Kelsen D, Ginsberg R, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Willett CG, Minsky BD. Longitudinal Quality-of-Life Analysis of RTOG 94-05 (Int 0123):A Phase III Trial of Definitive Chemoradiotherapy for Esophageal Cancer. Gastrointest Cancer Res. 2011 Mar;4(2):45-52. PMID 21673875
- [Result] Minsky BD, Pajak TF, Ginsberg RJ, Pisansky TM, Martenson J, Komaki R, Okawara G, Rosenthal SA, Kelsen DP. INT 0123 (Radiation Therapy Oncology Group 94-05) phase III trial of combined-modality therapy for esophageal cancer: high-dose versus standard-dose radiation therapy. J Clin Oncol. 2002 Mar 1;20(5):1167-74. doi: 10.1200/JCO.2002.20.5.1167. PMID 11870157
- [Result] Kachnic LA, Scott C, Ginsberg R, et al.: One year follow-up reveals no difference in quality of life between high dose and conventional dose radiation: a quality of life assessment of RTOG 94-05. [Abstract] Int J Radiat Oncol Biol Phys 51 (3 suppl 1): A-172, 97, 2001.
- [Result] Minsky BD, Berkey B, Kelsen DK, et al.: Preliminary results of Intergroup INT 0123 randomized trial of combined modality therapy (CMT) for esophagel cancer: standard vs high dose radiation therapy. [Abstract] Proceedings of the American Society of Clinical Oncology 19: A927, 2000.